CLINICAL TRIAL: NCT05617079
Title: The State of Nebulizer Therapy in Russian Federation: a National Survey Among Medicine Physicians
Brief Title: The State of Nebulizer Therapy in Russian Federation
Acronym: SoNeT
Status: Active, not recruiting | Type: Observational
Sponsor: Russian Federation of Anesthesiologists and Reanimatologists (Other)
Responsible Party: Sponsor
Other Study IDs: FARCT0004
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Survey; Respiratory Failure; Respiratory Disease
MeSH Terms: conditions — Respiratory Insufficiency; Respiration Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medicine physicians: Anesthesiologists, intensive care specialists, heads of departments of anesthesiology and intensive care, deputy chief physicians for anesthesiology and intensive care (heads of centers), employees of the department of anesthesiology and intensive care, pulmonologists working in medical organizations that use nebulizer therapy.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — an electronic survey will be conducted

SUMMARY:
It is known that the inhalation (nebulizer) use of drugs is of great importance in the intensive care of patients with acute and chronic respiratory failure of various origins.

Searching PubMed data for the last 5 years (2017-2022) for the keywords "nebulizer therapy" revealed 533 publications, and "mesh nebulizer therapy" - only 25 sources.

During the same period, the national database (E-Library) has 75 publications for the keywords "nebulizer therapy", and 4 sources for "mesh nebulizer therapy".

It should be noted that almost all publications are devoted to the use of nebulizers for specific diseases and pathological syndromes. There are no works evaluating the adherence of specialists, systemic indications and actually used methods.

The aim of trial is to study the current state of the use of nebulizer therapy in medical organizations and identify ways to improve its effectiveness This study is planned to be carried out using a questionnaire using a database based on the Internet electronic survey form.

DETAILED DESCRIPTION:
We intend to involve at least 3 medical organizations in the subjects of the Russian Federation with a population of up to 1 million people; at least 5 medical organizations in the constituent entities of the Russian Federation with a population level of 1 to 3 million people, at least 7 organizations with a population level of more than 3 million people. In cities of the Russian Federation with a population of 1 million people or more - at least 5 medical organizations, and in the cities of Moscow and St. Petersburg - at least 10 medical organizations.

ELIGIBILITY:
Inclusion Criteria:

* Medical physicians

Exclusion Criteria:

* Lack of experience in conducting nebulizer therapy. Lack of technical capability for nebulizer therapy in a medical organization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medicine physicians (VMP) practicing in the hospital and in the community settings.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Structure of indications, methods and frequency of use of nebulizer therapy | up to 1 month after inclusion
  Registration of the structure and indications for nebulizer therapy

SECONDARY OUTCOMES:
Drugs and frequency of their use during nebulizer therapy | up to 6 month after inclusion
  Registration of drugs used for nebulizer therapy
The frequency of use of nebulizer therapy for high-flow oxygen therapy, non-invasive ventilation and mechanical ventilation | up to 6 month after inclusion
  Frequency of use of nebulizer therapy for various types of respiratory support

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Gritsan, MD, Principal Investigator — Krasnoyarsk State Medical University n.a. prof. V.F. Voyno-Yasenetsky
Locations (1):
- Alexey Gritsan, Krasnoyarsk, Russia

IPD SHARING:
Plan to Share IPD: No